CLINICAL TRIAL: NCT05725928
Title: Randomized Trial of Assisted Ambulation to Improve Health Outcomes for Older Medical Inpatients
Brief Title: Assisted Ambulation to Improve Health Outcomes for Older Medical Inpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Michael Rothberg, Vice Chair for Research, Primary Care Institute, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 22-426; 1R01AG073278-01A1 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-02-13 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mobility Limitation; Frailty; Hospital Acquired Condition; Weakness, Muscle
MeSH Terms: conditions — Mobility Limitation; Frailty; Iatrogenic Disease; Muscle Weakness

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): No intervention
- Mobility Technician (Experimental): Designated mobility technicians (MT) will ambulate hospitalized medical patients up to 3 times daily, 7 days per week, until discharge or a maximum of 10 days. Each day, the MT will visit the patient 4 times or until the patient successfully ambulates 3 times that day. In cases where a PT has provided a recommendation in the patient's chart, the MT will follow the recommendation, if feasible. Otherwise, the MT will execute the standard mobility protocol. The mobility protocol will allow the MT to assist a patient with an appropriate out-of-bed activity based on their 6-clicks score from the immediately preceding session
  Interventions: Behavioral: Mobility technician

INTERVENTIONS:
Behavioral: Mobility technician — Designated mobility technicians (MT) will ambulate hospitalized medical patients up to 3 times daily, 7 days per week, until discharge or a maximum of 10 days. Each day, the MT will visit the patient 4 times or until the patient successfully ambulates 3 times that day. In cases where a PT has provided a recommendation in the patient's chart, the MT will follow the recommendation, if feasible. Otherwise, the MT will execute the standard mobility protocol. The mobility protocol will allow the MT to assist a patient with an appropriate out-of-bed activity based on their 6-clicks score from the immediately preceding session.
  Arms: Mobility Technician

SUMMARY:
The investigator proposes to conduct a randomized trial of supervised ambulation delivered by mobility technician (MT) up to three times daily, including weekends, to hospitalized medical patients. The aims of the study are to compare the short and intermediate-term outcomes of patients randomized to the intervention versus those patients randomized to receive usual care, to identify patients who are most likely to benefit from the intervention and to assess whether the intervention increases or decreases overall costs of an episode of care, including the cost of the MTs, the index hospitalization and the first 30 days post enrollment.

DETAILED DESCRIPTION:
The investigator proposes to conduct a large randomized trial to test the impact of MTs (Mobility Technicians) on short and intermediate term outcomes for 3000 patients aged 65 years and older at 5 hospitals in 2 health systems. Patients will be randomized to receive supervised ambulation up to 3 times daily with a MT or to receive usual care. All participants will wear an accelerometer on their wrist to track their movement throughout the hospital stay. The study has 3 aims. First, the study will compare the mobility of patients at discharge (or 10 days) to assess the impact of the MTs on this outcome. Of particular interest is whether the use of MTs will increase the proportion of patients who can go home vs.post-acute care, and whether the improvements in mobility are sustained at 30 days. Second, the study will use predictive modeling to identify which patients are most likely to benefit from this intervention. Third, the study will assess the impact of the intervention on overall costs associated with the episode of care, including inpatient costs and the 30 days post enrollment. This information will be important to convince health systems to adopt this approach.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria listed below to participate in this study:

1. ≥65 years of age
2. Admitted to a medical service
3. Complete history and physical examination on file
4. 6-Clicks score of 16-23
5. Insurance with Traditional Medicare or Medicare Advantage

Exclusion Criteria:

Any patient meeting any of the exclusion criteria listed below at baseline will be excluded from study participation:

1. Significant language barrier that requires a translator (other than Spanish at Baystate site only)
2. Discharge planned for that day or the following day
3. Observation status
4. Surgical procedure planned
5. Patients diagnosed with unstable angina or other medical conditions precluding participation in exercise/ambulation
6. Permanent residence in a skilled nursing facility
7. Comfort care measures only
8. >48 hours since admission
9. Active infection with COVID-19
10. Other active infection requiring contact or droplet precautions
11. Order for bedrest

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-10-11 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) from admission | Up to 10 days
  Every patient will have an SPPB score on admission to the study. A blinded assessor will measure the SPPB again at discharge or on day 10 if the patient is still hospitalized. The primary outcome is change from admission to discharge. Investigators will also compare the percentage of patients who reach the minimal clinically important difference of 1 point.
  SPPB minimum value= 0 SPPB maximum value= 12 (higher score indicates a better outcome). If no blinded team member is available, the evaluation may be carried out by any unblinded team member. The blinding status of the evaluator will be noted in REDCap.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) physical function - mobility | 30 days post enrollment
  Patients will complete the PROMIS physical function mobility bank via REDCap at 30 days post enrollment. PROMIS allows use of computer-adapted testing to measure patient-reported outcomes. The mobility question bank focuses on activities of physical mobility such as getting out of bed or a chair to walking up stairs. PROMIS measures were developed and validated with state-of-the-science methods supported by National Institutes of Health (NIH) funding. PROMIS was designed to enhance communication between clinicians and patients in diverse research and clinical settings and to be relevant across all conditions for the assessment of symptoms and functions.
  PROMIS minimum value= 0 PROMISE maximum value= 100 (higher score indicates a better outcome)
Activity Measure for Post-Acute Care (AM-PAC) basic mobility outpatient short form (SF) | 30 days post enrollment
  Subjects will complete the AM-PAC at 30 days post enrollment and the score will be transformed using the t-scale. In addition to comparing AM-PAC scores at 30 days, the investigator will also compare change in t-score from admission. The AM-PAC 6-clicks (assessed in the hospital) and the AM-PAC outpatient SF are normed to the same t-scale, allowing for conversion from the one to the other. The 6-clicks is scored by a clinical proxy, while the SF AM-PAC is self-reported, allowing for initial assessment by the MT and 30-day self-report by the patient. Previous studies have demonstrated adequate validity of mobility assessment via the AM-PAC using clinical or family proxies. To improve interpretability, investigators will compare the percentage of patients who reach the minimal clinically important difference of 3 points on the t-scale.
  AM-PAC minimum value= 29.41 AM-PAC maximum value= 80.30 (higher score indicates a better outcome)
Hospital-Acquired Complications | 10 days
  Composite outcome of venous thromboembolism, fall with injury, pressure ulcers or hospital-acquired pneumonia. Hospital-acquired complications will be identified from the electronic health record and from the falls reporting system. All falls will be examined, whether occurring during assisted ambulation or otherwise. Only falls with injury will be included in the hospital-acquired complications measure. Outcomes will be adjudicated by blinded reviewers. While investigators are primarily interested in the composite measure, investigators will also examine the individual components separately.
Number of Patients with Readmission within 30 days | 30 days after discharge
  All cause readmission within 30 days of discharge from the index hospitalization.
Activities of Daily Living | 30 days post enrollment
  Activities of daily living as measured by the Katz and Lawton scales.
  Katz minimum value= 0 Katz maximum value= 6 (higher score indicates a better outcome) Lawton minimum value= 0 Lawton maximum value= 8 (higher score indicates a better outcome)
Frailty | 30 days post enrollment
  Frailty as measured by the Fatigue, Resistance, Ambulation,Illness, and Loss of weight (FRAIL) scale.
  FRAIL minimum value= 0 FRAIL maximum value= 5 (higher score indicates a worse outcome)
Total episode cost | Admission to 30 days post enrollment
  Investigators will estimate total cost of the episode of care including the index admission (from hospital cost accounting systems), the personnel costs for the MTs (using hourly wages plus benefits), and all non-medication costs for the 30 days post-enrollment (from Medicare claims).
Number of Patients Discharged to Home | date of randomization to date of discharge, up to 30 days
  Based on the discharge disposition in the medical record, investigators will identify whether the patient was discharged to home.
Length of Stay | date of admission to date of discharge, up to 30 days
  Length of stay will be calculated as whole days from the time of admission to the time of discharge.
Mortality | 30 days from admission
  Patient's vital status will be ascertained from the EHR, Medicare claims or from follow-up phone calls.
Total episode cost | Admission to 6 months after enrollment
  Investigators will estimate total cost of the episode of care including the index admission (from hospital cost accounting systems), the personnel costs for the MTs (using hourly wages plus benefits), and all non-medication costs for the 6 months post-enrollment (from Medicare claims).
Falls post-discharge | 30 days from admission
  Whether the patient has fallen, whether it was multiple times and whether an injury occurred will be assessed via telephone
RCSQ (Richards Campbell Sleep Questionnaire) | Days 1-10
  Five question sleep survey which measures overall quality of sleep. Patients in both study arms will complete the questionnaire each morning regarding the previous night's sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rothberg, M.D., Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (5):
  - Baystate Medical Center, Springfield, Massachusetts
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic- Main Campus, Cleveland, Ohio
  - Marymount Hospital, Garfield Heights, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio

REFERENCES:
- [Background] Suter LG, Li SX, Grady JN, Lin Z, Wang Y, Bhat KR, Turkmani D, Spivack SB, Lindenauer PK, Merrill AR, Drye EE, Krumholz HM, Bernheim SM. National patterns of risk-standardized mortality and readmission after hospitalization for acute myocardial infarction, heart failure, and pneumonia: update on publicly reported outcomes measures based on the 2013 release. J Gen Intern Med. 2014 Oct;29(10):1333-40. doi: 10.1007/s11606-014-2862-5. Epub 2014 May 14. PMID 24825244
- [Background] Brown CJ, Roth DL, Allman RM, Sawyer P, Ritchie CS, Roseman JM. Trajectories of life-space mobility after hospitalization. Ann Intern Med. 2009 Mar 17;150(6):372-8. doi: 10.7326/0003-4819-150-6-200903170-00005. PMID 19293070
- [Background] Zisberg A, Shadmi E, Sinoff G, Gur-Yaish N, Srulovici E, Admi H. Low mobility during hospitalization and functional decline in older adults. J Am Geriatr Soc. 2011 Feb;59(2):266-73. doi: 10.1111/j.1532-5415.2010.03276.x. PMID 21314647
- [Background] Corcoran PJ. Use it or lose it--the hazards of bed rest and inactivity. West J Med. 1991 May;154(5):536-8. PMID 1866946
- [Background] Gillick MR, Serrell NA, Gillick LS. Adverse consequences of hospitalization in the elderly. Soc Sci Med. 1982;16(10):1033-8. doi: 10.1016/0277-9536(82)90175-7. PMID 6955965
- [Background] Hirsch CH, Sommers L, Olsen A, Mullen L, Winograd CH. The natural history of functional morbidity in hospitalized older patients. J Am Geriatr Soc. 1990 Dec;38(12):1296-303. doi: 10.1111/j.1532-5415.1990.tb03451.x. PMID 2123911
- [Background] Sager MA, Franke T, Inouye SK, Landefeld CS, Morgan TM, Rudberg MA, Sebens H, Winograd CH. Functional outcomes of acute medical illness and hospitalization in older persons. Arch Intern Med. 1996 Mar 25;156(6):645-52. PMID 8629876
- [Background] Brown CJ, Redden DT, Flood KL, Allman RM. The underrecognized epidemic of low mobility during hospitalization of older adults. J Am Geriatr Soc. 2009 Sep;57(9):1660-5. doi: 10.1111/j.1532-5415.2009.02393.x. Epub 2009 Aug 4. PMID 19682121
- [Background] Heit JA, Silverstein MD, Mohr DN, Petterson TM, O'Fallon WM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism: a population-based case-control study. Arch Intern Med. 2000 Mar 27;160(6):809-15. doi: 10.1001/archinte.160.6.809. PMID 10737280
- [Background] Campbell AJ, Borrie MJ, Spears GF. Risk factors for falls in a community-based prospective study of people 70 years and older. J Gerontol. 1989 Jul;44(4):M112-7. doi: 10.1093/geronj/44.4.m112. PMID 2738307
- [Background] Fisher SR, Kuo YF, Graham JE, Ottenbacher KJ, Ostir GV. Early ambulation and length of stay in older adults hospitalized for acute illness. Arch Intern Med. 2010 Nov 22;170(21):1942-3. doi: 10.1001/archinternmed.2010.422. No abstract available. PMID 21098357
- [Background] Graf C. Functional decline in hospitalized older adults. Am J Nurs. 2006 Jan;106(1):58-67, quiz 67-8. doi: 10.1097/00000446-200601000-00032. PMID 16481783
- [Derived] Johnson JK, Hamilton AC, Hu B, Pack QR, Lindenauer PK, Fox RJ, Hashmi A, Siegmund LA, Burchill CN, Taksler GB, Goto T, Stilphen M, Rothberg MB. Assisted ambulation to improve health outcomes for older medical inpatients (AMBULATE): study protocol for a randomized controlled trial. Trials. 2023 Jul 24;24(1):471. doi: 10.1186/s13063-023-07501-y. PMID 37488588